CLINICAL TRIAL: NCT01800279
Title: Comparative Study on the Effectiveness of Physical Therapy and Deontology for Temporomandibular Joint Dysfunction in Patients With Fibromyalgia Syndrome.
Brief Title: Physiotherapy and Deontology in the Temporomandibular Joint Dysfunction in Patients With Fibromyalgia Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Universidad de Granada (Other); Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UAL-12
Record Dates: First submitted 2013-02-19; First posted 2013-02-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Fibromyalgia Syndrome, Temporomandibular Joint, Pain.
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deontology Therapy (Active Comparator): The patients in the control group will port a deprogramming occlusal splint to sleep every night, an average of 8 hours per day, for 12 weeks of the treatment.
  Interventions: Other: Deontology Therapy
- Physiotherapy Protocol (Experimental): The physiotherapy protocol involves the application of kinesitherapy techniques and a myofascial therapy protocol. This protocol will be administered twice a week for 12 weeks.
  Interventions: Other: Physiotherapy Protocol

INTERVENTIONS:
Other: Physiotherapy Protocol — Kinesitherapy
  * Patient: supine position on the stretcher with a loop of 6 cm in the cervical area.
  * Tongue in the palate for all applied exercises.
  * Repetitions of each exercise: 8. Cervical traction. Cranium fore flexion 15 °. Open-close mouth dental contactless (10mm). Opening movement with a small resistor (one finger on chin).
  Flexion of the head, without actually lifting, resisting in the front. Occipital extension. Cranium fore flexion 15 °. Cervical traction.
  Myofascial Therapy. Induction suboccipital. Compression - decompression of the TMJ (Temporomandibular Joint). Horizontal Induction TMJ. Deep fascia induction in the temporal region. Deep Induction of the masseter fascia. Deep Induction of the external pterygoid. Induction of intraoral pterygoid.
  Arms: Physiotherapy Protocol
Other: Deontology Therapy — For the realization of the splint, the following protocol will be developed at the Faculty of Dentistry of Granada (Spain):
  * Impression of the maxilla with chromatic alginate "Phase plus" (Zhermack ©, Rovigo, Italy).
  * Emptying working models in plaster-stone type IV "Elite Rock" (Zhermack ©, Rovigo, Italy).
  * Deprogramming occlusal splints were made of polyester plates with terephthalic acid of 3 mm thick Clear 120 model (Dentaflux ©, Ripoll, Madrid). We used a molding machine of thermoplastic vacuum plate "The Machine" Dentaflux ©, Ripoll, Madrid.
  Arms: Deontology Therapy

SUMMARY:
The purpose of this study is to determine whether kinesitherapy techniques and a myofascial therapy protocol are effective in the treatment of temporomandibular joint dysfunction in patients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
Design: randomized clinical trial. Objective: to compare the therapeutic effects of physiotherapy and deontology protocol to improve pain, quality of life, physical function, quality of sleep, depression, anxiety, clinical severity, clinical improvement, and diagnostic criteria for research temporomandibular joint dysfunction in patients with fibromyalgia syndrome (FMS).

Background: the results on physiotherapy benefits for temporomandibular joint dysfunction in patients with FMS are controversial. Descriptive data and intervention studies are still scarce.

Methods and measures: sixty patients will be randomly assigned to experimental or control group. The experimental group will receive 24 sessions (twice a week) of kinesitherapy and myofascial release protocol, whereas the control group will undergo to deontology therapy (porting a deprogramming occlusal splint every night, an average of 8 hours per day, for 12 weeks of the treatment). Pain levels, impact of FMS symptoms, quality of sleep, depression, anxiety, clinical severity, clinical improvement and diagnostic criteria for research of temporomandibular joint dysfunction will be collected in both groups at baseline and 12 weeks after 48-hr the last intervention in the experimental and control groups, by an assessor blinded to the treatment allocation of the patients. Baseline demographic and clinical variables will be examined between both groups independent Student t-test for continuous data and χ2 tests of independence for categorical data. Separate 2x2 mixed model ANCOVAs with time (pre-post) as the within-subjects factor, group (experimental, control) will be to determine the effects of the treatment on pain, function, quality of sleep,depression, anxiety, clinical severity, clinical improvement and diagnostic criteria for research of temporomandibular joint dysfunction as the dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia syndrome.
* Agreement to attend evening therapy sessions.
* A chief complaint of acute pain (duration <6 months) in the temporomandibular joint on at least one side.
* The presence of joint clicking during jaw opening that was eliminated on protrusive opening.

Exclusion Criteria:

* History of recent trauma.
* Therapeutic co-interventions during treatment.
* Indication for surgical treatment of temporomandibular joint.
* Edentulism.
* Physical or mental illness that precludes attendance at therapy sessions.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | At baseline and 12 weeks
  The visual analog scale (VAS), designed to measure the intensity of pain and degree of relief experienced by the patient; with the value 0 for pain-free and 100 for maximum pain.

SECONDARY OUTCOMES:
Temporomandibular Dysfunction. | At baseline and 12 weeks
  Dworkin and LeResche present a multiaxial evaluation system that integrates the relevant aspects for the temporomandibular dysfunction in two axes. The exploration model consists of a protocol detailing the tests to be applied, and other specifications of the procedure to be followed by the professional:
  1. Temporomandibular pain.
  2. Pattern jaw opening.
  3. Vertical movement range.
  4. Sounds of the temporomandibular joint in palpation during vertical movement.
  5. Mandibular excursive movements.
  6. Pain extraoral muscle tenderness.
  7. Joint pain on palpation.
  8. Muscle pain during intraoral palpation.
Quality of Life (SF-36) | At baseline and 12 weeks
  The assessment of Quality of Life (SF-36) covers 8 dimensions of health status. It contains 36 items covering two areas, the functional status and the emotional wellness. The area of the functional state is represented by the following dimensions: physical function (10 items), social function (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items). The wellness area includes the dimensions of mental health (5 items), vitality (4 items), pain (2 items). Finally, the general health assessment includes the dimension of perception of general health (5 items) and the health change over the time (one item, which is not part of the final score).
Index of Widespread Pain and Symptom Severity | At baseline and 12 weeks
  This simple clinical case definition of fibromyalgia properly classifies the 88.1% of the cases classified by the ACR (American College of Rheumatology) classification criteria, and it does not require a physical or tender point. The symptom severity score allows the assessment of the severity of the symptoms of fibromyalgia in people with current or previous fibromyalgia, and those in which the criteria have not been applied yet. This questionnaire is especially useful in the longitudinal assessment of patients with marked symptom variability.
Physical Function. | At baseline and 12 weeks
  The fibromyalgia impact questionnaire (FIQ) consists of 10 items. The first item is composed of 11 subitems in which is valued the physical function. In the second and third items, patients indicate the number of days in which they disrupt their daily activity due to pain, or otherwise the days they find improvement. The impact caused by the symptoms of fibromyalgia in the physical and mental health of the patients was measured by the Spanish version of the Impact of Fibromyalgia Questionnaire. The FIQ assesses the following dimensions: feeling good, physical function, missing work and work capacity, physical, psychological and social components and global wellness. Also, it includes six visual analog scales for assessing fatigue, pain, stiffness, morning tiredness, anxiety and depression.
Quality of Sleep. | At baseline and 12 weeks
  Pittsburgh Sleep Quality Index Questionnaire (PSQI) consists of 24 items, and which interrogate issues such as the quality of sleep that the subject he has, or the frequency of certain events - such as difficulty falling asleep during the first half an hour or the presence of nightmares- are answered by an ordinal scale with four grades. In the correction of this questionnaire, seven scores are obtained which inform us of the components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, the use of hypnotic medication, and daytime dysfunction. Each of these components receives a discrete score which can range from 0 to 3. A score of 0 indicates that there are no problems in this respect, and a score of 3 indicates serious problems at that level. The sum of the scores in each partial component generates a total score, which can range from 0 to 21.
Rates of Depression | At baseline and 12 weeks
  The Beck inventory for depression is a self-administered questionnaire of 21 items that assesses a wide range of depressive symptoms. Its content emphasizes more the cognitive component of depression, and the symptoms of this area represent about 50% of the total score of the questionnaire, with symptoms of somatic / vegetative. In the second block, of the 21 items, 15 refer to eco-cognitive symptoms, and the remaining 6 to somatic-vegetative symptoms. Each item has four response alternatives listed from low to high severity, assessing the severity / intensity of the symptom. The range of the score is 0-63 points. The aim of this questionnaire is to quantify the symptoms, not provide a diagnosis. The breakpoints usually accepted to graduate the intensity/severity are the followings:
  * No Depression: 0-9 points.
  * Mild depression: 10-18 points
  * Moderate Depression: 19-29 points
  * Severe depression: ≥ 30 points
State-Trait Anxiety. | At baseline and 12 weeks
  The State-Trait Anxiety Inventory (STAI) measures a stable personality dimension (trait anxiety or tendency to anxiety), also includes a subscale of state, to detect anxiety behaviors. In the questionnaire, consisting of 40 items (20 for each level), the subjects have to describe how they feel generally, in the case of the trait anxiety scale, and how they feel when they answer, in the case of anxiety scale as a state. The STAI allows obtaining the scores of both scales separately.

OTHER OUTCOMES:
Clinical Impression of Severity. | At baseline and 12 weeks
  The clinical impression of severity scale assesses the severity level regarding the patient's physical condition. It comprises a Likert scale extending from a value of 1 (no disease) to a value of 7 (extremely ill).
Clinical Global Impression Improvement. | At baseline and 12 weeks
  The clinical global impression of improvement allows to evaluate the improvement perceived by the patient. It comprises a Likert scale which extends from a value of 1 (very much improved) to a value of 7 (extremely ill).

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida M Castro-Sánchez, PhD, Study Director — Universidad de Almeria
Locations (1):
- Fibromyalgia Association (AGRAFIM), Granada, Almeria, Spain

REFERENCES:
- [Background] Miernik M, Wieckiewicz M, Paradowska A, Wieckiewicz W. Massage therapy in myofascial TMD pain management. Adv Clin Exp Med. 2012 Sep-Oct;21(5):681-5. PMID 23356206
- [Background] de Felicio CM, Medeiros AP, de Oliveira Melchior M. Validity of the 'protocol of oro-facial myofunctional evaluation with scores' for young and adult subjects. J Oral Rehabil. 2012 Oct;39(10):744-53. doi: 10.1111/j.1365-2842.2012.02336.x. Epub 2012 Aug 1. PMID 22852833
- [Background] Guarda-Nardini L, Stecco A, Stecco C, Masiero S, Manfredini D. Myofascial pain of the jaw muscles: comparison of short-term effectiveness of botulinum toxin injections and fascial manipulation technique. Cranio. 2012 Apr;30(2):95-102. doi: 10.1179/crn.2012.014. PMID 22606852
- [Background] Richardson K, Gonzalez Y, Crow H, Sussman J. The effect of oral motor exercises on patients with myofascial pain of masticatory system. Case series report. N Y State Dent J. 2012 Jan;78(1):32-7. PMID 22474795
- [Background] Manfredini D, Castroflorio T, Perinetti G, Guarda-Nardini L. Dental occlusion, body posture and temporomandibular disorders: where we are now and where we are heading for. J Oral Rehabil. 2012 Jun;39(6):463-71. doi: 10.1111/j.1365-2842.2012.02291.x. Epub 2012 Mar 21. PMID 22435603
- [Background] Aggarwal A, Keluskar V. Physiotherapy as an adjuvant therapy for treatment of TMJ disorders. Gen Dent. 2012 Mar-Apr;60(2):e119-22. PMID 22414516
- [Background] Walczynska-Dragon K, Baron S. The biomechanical and functional relationship between temporomandibular dysfunction and cervical spine pain. Acta Bioeng Biomech. 2011;13(4):93-8. PMID 22339095
- [Background] Craane B, Dijkstra PU, Stappaerts K, De Laat A. Randomized controlled trial on physical therapy for TMJ closed lock. J Dent Res. 2012 Apr;91(4):364-9. doi: 10.1177/0022034512438275. Epub 2012 Feb 8. PMID 22318373
- [Background] Dym H, Israel H. Diagnosis and treatment of temporomandibular disorders. Dent Clin North Am. 2012 Jan;56(1):149-61, ix. doi: 10.1016/j.cden.2011.08.002. PMID 22117948
- [Background] Doepel M, Nilner M, Ekberg E, LE Bell Y. Long-term effectiveness of a prefabricated oral appliance for myofascial pain. J Oral Rehabil. 2012 Apr;39(4):252-60. doi: 10.1111/j.1365-2842.2011.02261.x. Epub 2011 Oct 11. PMID 21985440
- [Background] Hunter EK. Integration of rehabilitation and acupuncture in the treatment of a professional musician with temporomandibular joint dysfunction. Acupunct Med. 2011 Dec;29(4):298-301. doi: 10.1136/aim.2010.003889. Epub 2011 Jun 16. PMID 21685109
- [Background] Armijo-Olivo S, Silvestre R, Fuentes J, da Costa BR, Gadotti IC, Warren S, Major PW, Thie NM, Magee DJ. Electromyographic activity of the cervical flexor muscles in patients with temporomandibular disorders while performing the craniocervical flexion test: a cross-sectional study. Phys Ther. 2011 Aug;91(8):1184-97. doi: 10.2522/ptj.20100233. Epub 2011 Jun 9. PMID 21659465
- [Background] Cuccia AM, Caradonna C, Caradonna D. Manual therapy of the mandibular accessory ligaments for the management of temporomandibular joint disorders. J Am Osteopath Assoc. 2011 Feb;111(2):102-12. PMID 21357496
- [Background] Ariji Y, Katsumata A, Hiraiwa Y, Izumi M, Sakuma S, Shimizu M, Kurita K, Ariji E. Masseter muscle sonographic features as indices for evaluating efficacy of massage treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Oct;110(4):517-26. doi: 10.1016/j.tripleo.2010.05.003. PMID 20868996
- [Background] Silant'eva EN. [The role of therapeutic exercises in the combined treatment and rehabilitation of patients with pain syndrome associated with the dysfunction of temporomandibular joint]. Vopr Kurortol Fizioter Lech Fiz Kult. 2010 May-Jun;(3):22-6. Russian. PMID 20737707
- [Background] La Touche R, Paris-Alemany A, von Piekartz H, Mannheimer JS, Fernandez-Carnero J, Rocabado M. The influence of cranio-cervical posture on maximal mouth opening and pressure pain threshold in patients with myofascial temporomandibular pain disorders. Clin J Pain. 2011 Jan;27(1):48-55. doi: 10.1097/AJP.0b013e3181edc157. PMID 20733480
- [Background] Santos Tde S, Piva MR, Ribeiro MH, Antunes AA, Melo AR, Silva ED. Lasertherapy efficacy in temporomandibular disorders: control study. Braz J Otorhinolaryngol. 2010 May-Jun;76(3):294-9. doi: 10.1590/S1808-86942010000300004. PMID 20658006
- [Background] Oliveira-Campelo NM, Rubens-Rebelatto J, Marti N-Vallejo FJ, Alburquerque-Sendi N F, Fernandez-de-Las-Penas C. The immediate effects of atlanto-occipital joint manipulation and suboccipital muscle inhibition technique on active mouth opening and pressure pain sensitivity over latent myofascial trigger points in the masticatory muscles. J Orthop Sports Phys Ther. 2010 May;40(5):310-7. doi: 10.2519/jospt.2010.3257. PMID 20436241
- [Background] Fricton JR, Ouyang W, Nixdorf DR, Schiffman EL, Velly AM, Look JO. Critical appraisal of methods used in randomized controlled trials of treatments for temporomandibular disorders. J Orofac Pain. 2010 Spring;24(2):139-51. PMID 20401352
- [Background] Fernandez-Carnero J, La Touche R, Ortega-Santiago R, Galan-del-Rio F, Pesquera J, Ge HY, Fernandez-de-Las-Penas C. Short-term effects of dry needling of active myofascial trigger points in the masseter muscle in patients with temporomandibular disorders. J Orofac Pain. 2010 Winter;24(1):106-12. PMID 20213036